CLINICAL TRIAL: NCT03322735
Title: A Study of BCMA CAR-T Cells for Patients With Relapse and Refractory Multiple Myeloma
Brief Title: Study of BCMA CAR-T in Multiple Myeloma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: The Pregene (ShenZhen) Biotechnology Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HenanCH284
Record Dates: First submitted 2017-10-19; First posted 2017-10-26 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-tumor response of BCMA CAR-T (Experimental): Drug: Cyclophosphamide patients will receive a standard pre-conditioning regime with cyclophosphamide 0.6-0.8g/m2/day IV for 2 days.
  Drug: Fludarabine Fludarabine 25-30mg/m2/day IV for 3 days. Biological: BCMA CAR-T BCMA CAR-T cells will be administered after completion of the chemotherapy.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: BCMA CAR-T

INTERVENTIONS:
Drug: Fludarabine — 25-30mg/m2/day IV for 3 days
Drug: Cyclophosphamide — cyclophosphamide 0.6-0.8g/m2/day IV for 2 days
Biological: BCMA CAR-T — BCMA CAR-T cells will be administered after completion of the chemotherapy.

SUMMARY:
The purpose of this study is to infusion BCMA CAR-T cells to the patients with relapsed and refractory multiple myeloma(MM), to assess the safety and feasibility of this strategy. The CAR enables the T cell to recognize and kill the MM cells through the recognition of BCMA, a protein expressed of the surface of the malignant plasma cells in MM patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 years to 70 years, expected survival > 3 months;
* 2. Confirmed diagnosis of active MM as defined by IMWG. BCMA expression of the malignant cells must be detected by immunohistochemistry or by flow cytometry.
* 3. BCMA-expressing B cell malignancy must be assured and must be relapsed or refractory disease.；
* 4. ECOG performance status of 0-2;
* 5. Cardiac function: 1-2 levels; Liver: TBIL≤3ULN，AST ≤2.5ULN，ALT ≤2.5ULN; kidney: Cr≤1.25ULN;
* 6. No serious allergic constitution;
* 7. No other serous diseases that conflicts with the clinical program;
* 8. No other cancer history;
* 9. female participants of reproductive potential must have a negative serum pregnancy test;
* 10. Subjects must have signed written, informed consent.

Exclusion Criteria:

* 1. Pregnant or lactating women;
* 2. Uncontrolled active infection, HIV infection, syphilis serology reaction positive;
* 3. Active hepatitis B or hepatitis C infection;
* 4. Recent or current use of glucocorticoid or other immunosuppressor;
* 5. serious mental disorder;
* 6. With severe cardiac, liver, renal insufficiency, diabetes and other diseases;
* 7. Participate in other clinical research in the past three months; previously treatment with any gene therapy products;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-12-08 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 1 year
  number of participants with adverse events

SECONDARY OUTCOMES:
Persistence of the BCMA CAR+ T cells | 1 year
  determine duration of in vivo survival of BCMA CAR-T cells
anti-tumor responses of BCMA CAR-T cells | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yongping Song, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Cancer Hospital Affiliate to Zhengzhou University & Henan Cancer Hospital, Zhengzhou, Henan, China